CLINICAL TRIAL: NCT04401826
Title: Evaluation of Pain Following Microsurgical Esthetic Crown Lengthening Using Flap Vs. Flapless Piezo-surgical Approach: A Randomized Controlled Clinical Trial
Brief Title: Micro-surgical Treatment of Gummy Smile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marie-line Sherif Sourour, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PER3-3-1
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The conventional approach (Experimental): Conventionnal ECL using piezosurgery and microsurgical tools
  Interventions: Procedure: Micro-surgical crown lengthening approach using Piezosurgery
- The intervention approach: (Active Comparator): Conventionnal ECL with tunneling using piezosurgery and microsurgical tools
  Interventions: Procedure: Tunneling micro-surgical crown lengthening approach using piezo-surgery

INTERVENTIONS:
Procedure: Tunneling micro-surgical crown lengthening approach using piezo-surgery — excess gingiva is eliminated. 2 mm bone is removed from CEJ-bone crest with piezo surgery via tunneling
  Arms: The intervention approach:
Procedure: Micro-surgical crown lengthening approach using Piezosurgery — excess gingiva is eliminated. 2 mm bone is removed from CEJ-bone crest with piezo surgery with conventional flap elevation.
  Arms: The conventional approach

SUMMARY:
Compare pain response following microsurgical conventional flap approach using Piezosurgery versus flapless approach for esthetic crown lengthening in management of patients with short clinical crowns in the upper anterior region.

DETAILED DESCRIPTION:
The conventional approach: Anesthesia will be given followed by bone sounding using William graduated periodontal probe and measuring the pocket depth (using magnification loupes and microsurgical blades)

* Marking the bleeding points
* An internal bevel incision is made followed afterwards by a sulcular incision.
* The gingival collar is eliminated.
* Elevation of the flap is proceeded to allow access for osteoplasty using piezo surgery and an apical position of the bone 2-3mm beyond CEJ.
* Mattress suture (6.0) is made

The intervention approach:

Surgery is done the same as in the conventional approach but without opening a flap, gaining access via a tunneling instrument and piezo tips for osteoplasty

ELIGIBILITY:
Inclusion Criteria:

1. Patients with healthy systemic condition.
2. Adult patients ˃ 18 years old.
3. The presence of the six upper anterior teeth.
4. Patients who have short clinical crowns due to altered passive eruption classified as Type I subclass B (Coslet, Vanarsdall and Weisgold, 1977).
5. Absence of sites with attachment loss and probing depth (PD) >3 mm.
6. Keratinized gingiva of at least 2mm width (Pontoriero and Carnevale, 2001).
7. Compliance with good oral hygiene.
8. Patients accepts 6-months follow-up period (cooperative patients).
9. Patients provides an informed consent.

Exclusion Criteria:

1. Presence of prosthetic crowns
2. Extensive restorations
3. Extensive incisal edge attrition.
4. Smokers ˃ 10 cigarettes / day
5. Pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-06 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Pain VAS | 48 hours
  Visual Analogue Scale for Pain (numbers from 0 to 10 ('no pain' to 'worst pain imaginable') measured daily for the first 2 days postoperative

SECONDARY OUTCOMES:
Mid-buccal gingival margin level | 6 months
  Periodontal probe with William's graduation will be used to measure the distance from a prefabricated grooved stent vertically- to the level of the gingival margin at the mid-buccal surface (measured at baseline, 3 and 6 months postoperatively)
Post-Surgical Patient Satisfaction. | 6 months
  Numerical Rating Scale (A 3-item questionnaire is asked, and the patients shall use a 7-point answer scale. )
Pink Esthetic Score | 6 months
  The PES is based on seven variables:
  mesial papilla, distal papilla, soft-tissue level, soft tissue contour, alveolar process deficiency, soft-tissue color and texture. Each variable shall be assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score. The mesial and distal papilla will be evaluated for completeness, incompleteness or absence. All other variables will be assessed by comparison to a reference tooth.
Post-Surgical swelling | 14 days
  Absent: no swelling, Slight: intraoral swelling at the operated area, Moderate: moderate intraoral swelling at the operated area and Intense: intensive extra oral swelling extending beyond the operated area. (Assessed in day 7 and 14 postoperatively)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medecine-CU, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No